CLINICAL TRIAL: NCT01240356
Title: Combined Lysis of Thrombus in Brain Ischemia With Transcranial Ultrasound and Systemic T-PA-Hands-Free. A Phase I/II Pilot Safety Trial
Brief Title: CLOTBUST Hands-Free: A Phase I/II Pilot Safety Trial
Acronym: CLOTBUST-HF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Grotta, MD, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOTBUST-HF
Record Dates: First submitted 2010-11-08; First posted 2010-11-15 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: transcranial doppler; sonothrombolysis; ultrasound; stroke
MeSH Terms: conditions — Stroke | interventions — Ultrasonography, Doppler, Transcranial; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I: Healthy Volunteers (Experimental): Subjects without history of Central Nervous System Disease will receive 2-hours of hands-free 2-megahertz (MHz) transcranial Doppler ultrasound insonation continuously. A brain MRI with gadolinium will be performed before and after the ultrasound.
  Interventions: Device: 2-MHz transcranial Doppler ultrasound
- Phase II: 0-3 hour Patients (Experimental): Ischemic stroke patients who present between 0-3 hours will receive 2-hours of hands-free 2-MHz transcranial Doppler ultrasound Continuously to the intracranial vessels.
  Interventions: Device: 2-MHz transcranial Doppler ultrasound insonation

INTERVENTIONS:
Device: 2-MHz transcranial Doppler ultrasound — 2-hours of hands-free ultrasound will be insonated continuously. A brain MRI with gadolinium will be performed before and after the ultrasound.
  Other Names: transcranial Doppler Ultrasound; ultrasound
  Arms: Phase I: Healthy Volunteers
Device: 2-MHz transcranial Doppler ultrasound insonation — 2-hours of hands-free ultrasound delivered to in the intracranial vessels.
  Other Names: transcranial Doppler ultrasound; ultrasound; sonothrombolysis
  Arms: Phase II: 0-3 hour Patients

SUMMARY:
The purpose of CLOTBUST-HF is to determine the safety of a novel, external Hands-Free transcranial Doppler (TCD) ultrasound system in healthy volunteers and ischemic stroke patients. If found to be safe, the widespread use of operator-independent, ultrasound-enhanced thrombolysis will allow the planning for a large Phase III efficacy trial.

DETAILED DESCRIPTION:
Ultrasound energy to enhance intravenous rt-PA thrombolysis is a promising novel treatment modality for ischemic stroke. Despite encouraging safety data utilizing diagnostic frequencies of transcranial Doppler (TCD) ultrasound, lack of widespread availability of trained personnel has limited its application.

- The primary specific aim for this pilot phase I/II study is to assess the safety of a novel, external Hands-Free TCD ultrasound system. Safety of the new Hands-Free TCD system will first be assessed in healthy volunteers. Safety in these participants will be determined by detailed neurological and dermatological exams and MRI imaging of the brain. Next, safety of the device will be evaluated in two distinct sets of acute ischemic stroke patients: 0-3 hour patients treated with standard IV rt-PA and 3-6 hour non-lytic, image-selected patients treated with sonolysis (with or without intravenous microbubbles). Among the healthy volunteers the primary measures of safety will be to have no detectable changes in a detailed neurological exam nor any blood- brain barrier (BBB) disruption or changes in permeability. Among both the 0-3 hour and 3-6 hour groups the primary measure of safety will be to not tolerate greater than a 10% rate of symptomatic intracerebral hemorrhage (sICH) within 24 hours.

* The primary hypothesis is that replacing conventional TCD ultrasound hand-held TCD technology with a Hands-Free system will be safe in healthy volunteers as well as acute ischemic stroke patients.

If the device is found to be safe in either the 0-3 hour or 3-6 hour groups,

- the secondary aims for this study will explore the rates of arterial recanalization in the 0-3 hour and/or 3-6 hour groups, favorable outcomes, and clinical recovery. The secondary aims will assess the hypothesis is that Hands-Free TCD will display similar recanalization and early clinical recovery rates compared to available historical diagnostic TCD ultrasound controls exposed to conventional FDA-approved TCD technology.

Data generated during this phase I/II trial will evaluate the safety of replacing an operator-dependent TCD device with an operator-independent unit. In turn, this will allow extensive availability of therapeutic ultrasound and improve enrollment into ultrasound-enhanced thrombolysis stroke trials.

ELIGIBILITY:
INCLUSION CRITERIA:

Phase I Safety (healthy volunteers):

* Presence of temporal windows as measured first by an FDA-approved diagnostic TCD device.
* Age ≥ 18 years old.
* Signed informed consent.

Phase II (0-3 hours ischemic stroke patients):

* Disabling focal neurological deficit (NIHSS > 4 points);
* No evidence of hemorrhage on non-contrast head CT scan;
* Intravenous rt-PA (0.9 mg/kg, 10% bolus 90% infusion over 1 hour, maximum dose 90 mg) infusion initiated within 3 hours of symptom onset;
* Diagnostic TCD completed and HF-TCD placed before rt-PA bolus.
* Diagnostic TCD confirms intracranial arterial occlusion of the middle cerebral artery (MCA), anterior cerebral artery (ACA), internal carotid artery (ICA), posterior cerebral artery (PCA) or distal basilar artery.
* Age ≥ 18 years old.
* Signed informed consent.

Phase II (3-6 hours ischemic stroke patients):

* Measurable focal neurological deficit (NIHSS > 4 points);
* No evidence of hemorrhage on non-contrast head CT scan;
* Diagnostic TCD confirms intracranial arterial occlusion of the middle cerebral artery (MCA), anterior cerebral artery (ACA), internal carotid artery (ICA), posterior cerebral artery (PCA) or distal basilar artery.
* Presence of neuroimaging defined mismatch (CT or MRI prior to enrollment)

  1. CT-perfusion

     * ≥ 20% difference between affected territories on Time to Peak (TTP) and Cerebral Blood Volume (CBV) maps.
  2. MRI Diffusion-Perfusion mismatch

     * ≥ 20% difference between diffusion-weighted imaging (DWI) lesion and territory of perfusion delay perfusion weighted imaging (PWI).
* Age ≥ 18 years old.
* Signed informed consent.

EXCLUSION CRITERIA:

Phase I Safety (healthy volunteers):

* History of any neurological disease affecting the central nervous system;
* Lack of temporal windows.
* History of renal disease or glomerular filtration rate (GFR) < 60.
* Contraindication to MRI (e.g., pacemaker, spinal cord stimulator, severe claustrophobia)

Phase II (0-3 hours ischemic stroke patients):

* Absent temporal windows in patients with anterior circulation ischemia;
* Intra-arterial thrombolysis;
* Patient refusal to give informed consent to participate in the CLOTBUST-HF trial;
* Contraindications for intravenous rt-PA (NINDS rt-PA Stroke Study Protocol)2.
* Phase II (3-6 hours ischemic stroke patients):
* Absent temporal windows in patients with anterior circulation ischemia;
* Intra-arterial thrombolysis;
* Patient refusal to give informed consent to participate in the CLOTBUST-HF trial;
* History of allergic response to Definity® microspheres or microbubbles currently being tested (MRX-801);
* Baseline imaging consistent with a malignant ischemic pattern (low CBV values or DWI territory >100cc of tissue);
* Baseline MRI imaging demonstrating delayed perfusion of > 8 seconds in >100cc of brain parenchyma26;
* Patients receiving other investigational drugs, procedures, or therapies within 30 days prior to study treatment;
* Significant concurrent medical/neurological conditions or deviation from normal laboratory test values at baseline that, in the opinion of the investigator, pose significant risk to the patient and warrant exclusion from the study;
* Known severe chronic obstructive pulmonary disease (COPD) (baseline oxygen saturation < 80% on room air);
* Known right-to-left cardiac shunt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Grotta, MD, Principal Investigator — UT Medical School-Houston
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UT Medical School-Houston, Houston, Texas

REFERENCES:
- [Result] Barlinn K, Barreto AD, Sisson A, Liebeskind DS, Schafer ME, Alleman J, Zhao L, Shen L, Cava LF, Rahbar MH, Grotta JC, Alexandrov AV. CLOTBUST-hands free: initial safety testing of a novel operator-independent ultrasound device in stroke-free volunteers. Stroke. 2013 Jun;44(6):1641-6. doi: 10.1161/STROKEAHA.113.001122. Epub 2013 Apr 18. PMID 23598523
- [Result] Barreto AD, Alexandrov AV, Shen L, Sisson A, Bursaw AW, Sahota P, Peng H, Ardjomand-Hessabi M, Pandurengan R, Rahbar MH, Barlinn K, Indupuru H, Gonzales NR, Savitz SI, Grotta JC. CLOTBUST-Hands Free: pilot safety study of a novel operator-independent ultrasound device in patients with acute ischemic stroke. Stroke. 2013 Dec;44(12):3376-81. doi: 10.1161/STROKEAHA.113.002713. Epub 2013 Oct 24. PMID 24159060
- [Derived] Al-hussain F, Hussain MS, Molina C, Uchino K, Shuaib A, Demchuk AM, Alexandrov AV, Saqqur M; CLOTBUST Investigators. Does the sex of acute stroke patients influence the effectiveness of rt-PA? BMC Neurol. 2014 Mar 26;14:60. doi: 10.1186/1471-2377-14-60. PMID 24669960

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Non-stroke volunteers.
- Phase II: Acute Ischemic Stroke patients received standard-doce intravenous tissue-type plasminogen activator (tPA) within 0-3 hours window.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 18 | 20
Completed | 15 | 20
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — MRI contraindication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Phase II-20 patients with ischemic stroke treated with IV-tPA
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 15 | 20 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 2 | 8 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16) | 63 (14) | 57 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  United States | 15 | 20 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase I Group With Blood-brain-barrier Disruption (BBB) as Measured by MRI of the Brain
Description: Phase I : Imaging of the brain via MRI scans was performed to determine if the Hands-Free transcranial Doppler (TCD) system results in any BBB-disruption or deterioration in permeability.
Time Frame: 2-3 hours after treatment
Measure: Number; unit: participants
Groups:
- Phase I: Non stroke patients
Arm/Group | Phase I
Number analyzed (Participants) | 15
participants | 0

2. Primary Outcome: Safety in Phase II Group as Measured by Incidence of Symptomatic Intracerebral Hemorrhage
Description: Phase II: Determine if the Hands-Free TCD will not result in higher than 10% rate of symptomatic intracerebral hemorrhage (ICH) within 24 hours (defined as clinical worsening > 4 NIH Stroke Scale (NIHSS) points and presence of hemorrhage on CT scan that in the opinion of the treating physician is causatively related to ICH on CT) in 0-3 hours acute stroke patients treated with intravenous tissue-type plasminogen activator (IV-t-PA).
Time Frame: within 24 hours
Population: Intention to Treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase II - Ischemic Stroke Patients: Phase II - A group of 20 patients with ischemic stroke treated with IV-tPA
Arm/Group | Phase II - Ischemic Stroke Patients
Number analyzed (Participants) | 20
percentage of patients | 0 [0 to 17]

3. Secondary Outcome: Number of Participants in Phase I Group With Adverse Events During and After Study Treatment With HF TCD
Description: Phase I - A group of healthy volunteers will be assessed to determine the feasibility and activity of hands-free (HF) transcranial Doppler (TCD). Adverse events include subject complaints regarding discomfort of the device and dermatological adverse events as evidenced by a detailed physical examination of skin integrity post-insonation.
Time Frame: 2-3 hours after treatment
Population: ITT
Measure: Number; unit: participants
Groups:
- Phase 1 (Healthy Volunteers): Phase I - A group of non-stroke healthy volunteers.
Arm/Group | Phase 1 (Healthy Volunteers)
Number analyzed (Participants) | 15
participants | 0

4. Secondary Outcome: Percentage of Participants in the Phase II Group That Show Arterial Recanalization as Measured Using Standard Transcranial Doppler Ultrasound Systems
Description: Ischemic stroke patients: 2-hour rates of arterial complete and partial recanalization as measured using standard Transcranial Doppler Ultrasound systems.
Time Frame: 2-3 hours after treatment
Population: ITT - Percent of patients who had complete recanalization after treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase II - Iscehmic Stroke Patients: Phase II - 20 patients with ischemic stroke treated with IV-tPA
Arm/Group | Phase II - Iscehmic Stroke Patients
Number analyzed (Participants) | 20
percentage of patients | 40 [19 to 64]

5. Secondary Outcome: Percentage of Participants in Phase II Group With Neurological Worsening as Determined by the NIH Stroke Scale
Description: The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. Each item on the NIHSS scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Time Frame: within 90 days of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase II - Ischemic Stroke Patients
Number analyzed (Participants) | 20
percentage of patients | 5 [0 to 25]

6. Secondary Outcome: Percentage of Participants in Phase II Group With Excellent Outcome as Measured by Modified Rankin Scale (mRS)
Description: A modified Rankin Scale (mRS) score of 0 or 1 indicates an excellent outcome. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The mRS scale ranks patients from 0 to 6 (0 is the best score, 6 is the worst score).
Time Frame: at 3-months from enrollment
Population: ITT with modified Ranking scores (mSR) at 90 days. % displayed is % with excellent outcome (mRS of 0-1).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase II - Ischemic Stroke Patients
Number analyzed (Participants) | 20
percentage of patients | 25 [7 to 49]

7. Primary Outcome: Number of Participants in Phase I Group With Neurological Deterioration as Measured by Neurological Examination
Description: The neurological examinations comprised assessments of mental status and orientation, cranial nerve examination, muscle strength and tone, deep tendon reflexes, sensory testing, coordination, and gait.
Time Frame: 2-3 hours after treatment
Measure: Number; unit: participants
Groups:
- Phase I: Healthy Volunteers: Phase I - A group of 15 Non-stroke healthy volunteers.
Arm/Group | Phase I: Healthy Volunteers
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Groups:
- Phase I: Healthy Volunteers: Phase I - 15 non-stroke healthy volunteers.
- Phase II - Ischemic Stroke Patients: Phase II - 20 patient with ischemic stroke treated with IV-tPA
Arm/Group | Phase I: Healthy Volunteers | Phase II - Ischemic Stroke Patients
Serious Adverse Events (participants affected / at risk) | 0/15 | 9/20
Other Adverse Events (participants affected / at risk) | 0/15 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Healthy Volunteers (N=15) | Phase II - Ischemic Stroke Patients (N=20)
Intracranial hemohhrage secondary to bacterial endocarditis (Nervous system disorders) | 0 (0) | 1 (1)
Death (Nervous system disorders) | 0 (0) | 3 (3)
Cerebral edema (Nervous system disorders) | 0 (0) | 4 (4)
Pneumonia/respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke progression/Nuero-worsening (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Healthy Volunteers (N=15) | Phase II - Ischemic Stroke Patients (N=20)
Fewer (Infections and infestations) | 0 (0) | 6 (6)
Anemia/decreased hemoglobin and hematocrit (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Hypertension (Cardiac disorders) | 0 (0) | 6 (6)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Electrolyze imbalance (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Right lung atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated CK (Cardiac disorders) | 0 (0) | 1 (1)
Elevated white blood count (Infections and infestations) | 0 (0) | 5 (5)
Utinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Asymptomatic ICH (Nervous system disorders) | 0 (0) | 6 (6)
Elevated Coag lab test (Nervous system disorders) | 0 (0) | 1 (1)
New diagnosis of PFO (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Positive sputum culture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The last phase (Phase II: 3-6 hour non-lytic patients who presented between 3-6 hours and with evidence of mismatch on neuroimaging), was not completed. This portion of the study was not started as new published evidence suggested little value.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes